CLINICAL TRIAL: NCT04026802
Title: Safety and Feasibility of a Novel In--Bed Resistance Training Device in Elderly Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-01905
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Old Age; Debility
Keywords: deconditioning of elderly inpatients; loss of functionality
MeSH Terms: conditions — Frailty | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In--Bed Resistance Training Device (Experimental): The present invention provides full body resistance training devices that attach to a planar edge, such as a footboard, headboard, or sideboard of a bed. The devices employ resistance bands for resistance training in both the incursion (force applying) and excursion (force releasing) phase of exercise.
  Interventions: Other: In-Bed Resistance Training Device
- Standard of Care (Active Comparator): No resistance training device
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: In-Bed Resistance Training Device — Physical Therapy using the in bed training device
  Arms: In--Bed Resistance Training Device
Other: Standard of Care — Does not include early implementation of physical therapy
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to decrease deconditioning of elderly inpatients in acute care institutions and to assess the safety and feasibility of a newly developed resistance training device. Investigators believe this device will help hospitalized seniors maintain their independence by preventing the loss of functionality from deconditioning and improve value of care through decreased length of stay and utilization of care. Current therapy will be complemented with a new in--bed resistance training device to target weak elderly patients and standardize progressive resistance training in facilities.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 70 years old
* Admitted to acute inpatient medicine unit at NYU Langone Health (17E and 17W) from - - - - - Emergency Department
* Receiving Physical Therapy
* Initial AMPAC 6 clicks score 11-18
* English Speaking

Exclusion Criteria:

* ICU level care
* Acute cardiac risk (including recent acute MI and stroke, unstable arrhythmias, or uncontrolled hypertension)
* Exercise-limiting physical disability (ie rotator cuff injury, neurologic impairment)
* Severe cognitive impairment (1) No significant dementia or delirium (2) Patient able to accept readiness for PT and comprehend education
* Contact Precautions

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
AMPAC 6 Clicks Composite PT (range 11-18) | 1 Year
  The AM - PAC measures 3 functional domains: basic mobility, daily activities and applied cognition . It may be used for assessment in adults with a wide range of diagnoses and levels of performance in the 3 domains . The '6 - Clicks' instruments may have advantages over the instruments previously developed for the acute care setting in that they are simple and quick to complete, provide a transparent measure of patients' capabilities in functional areas important for prioritization of therapy resources , and use Item Response Theory to derive a common metric that can be linked with other short forms derived from the AM - PAC instrument.

SECONDARY OUTCOMES:
Grip Strength using a dynamometer | 30 seconds
  Quantified by measuring the amount of static force that the hand can squeeze around a dynamometer
Modified 30 second sit to stand | 1 Year
  Count of the number of times a patient is able to come to a modified standing position in 30 seconds
SF-12 | 1 Year
  Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Moroz, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States